CLINICAL TRIAL: NCT05643352
Title: Patient-reported Outcomes of Barbed Reposition Pharyngoplasty in Unilevel Palatal Snoring: a Prospective Study
Brief Title: Barbed Reposition Pharyngoplasty in Patients Complaining of Unilevel Palatal Snoring
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AZ Delta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18059
Record Dates: First submitted 2022-11-23; First posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Snoring; Sleep-Disordered Breathing
Keywords: Pharyngoplasty; Barbed reposition pharyngoplasty; Snoring; Surgery
MeSH Terms: conditions — Snoring; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Barbed reposition pharyngoplasty — Barbed reposition pharyngoplasty was performed in all patients

SUMMARY:
The aim of the study is to determine whether there is a statistically significant difference in snoring intensity before and after performing a Barbed Reposition Pharyngoplasty as a single-level snoring procedure. The investigators aim to determine whether this is a valid alternative to the more classical techniques of pharyngoplasty. Furthermore, the investigators also wish to map the various postoperative complications and compare them with those of the more conventional techniques. The investigators compare the snoring intensity before surgery with the snoring intensity at 2 weeks (first postoperative control), at 6 weeks (second postoperative control) and at 6 months (Third postoperative control).

For the evaluation of snoring, the investigators use 4 scales/questionnaires. These questionnaires are currently also used as standard at the outpatient clinic for snoring problems. These 4 scales/questionnaires are completed at every check-up.

During the first postoperative check-up, the postoperative side effects are checked (bleeding, infection, readmission, needed consultation with another doctor, date of resumption of work). The investigators also map the pain with a visual analog scale and measure this the day after the operation and let the patient fill it in 3 days, 1 week and 2 weeks after the operation.

ELIGIBILITY:
Inclusion Criteria:

* single-level retro-palatal collapse observed during drug-induced sleep endoscopy (DISE)

Exclusion Criteria:

* OSAS defined as having an obstructive AHI (OAHI) ≥ 30
* Obese patients with a body mass index (BMI) ≥ 30 kg/m².
* Patients with multilevel airway collapse observed during DISE
* Patients younger than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Change in Snoring intensity | At 2 weeks, at 6 weeks and at 6 months
  Seld-reported subjective score from 0 to 10 that describes the impact of snoring with 0 meaning no snoring and 10 meaning sleeping separately from partner
Change in Snoring severity | At 2 weeks, at 6 weeks and at 6 months
  Seld-reported subjective score that describes the severity of snoring (frequency, duration,...). Score from 0 to 9 with 0 meaning never snoring and 9 meaning snoring every night during the entire night with sounds audible from another floor
Change in Snoring score | At 2 weeks, at 6 weeks and at 6 months
  Seld-reported subjective score that describes the overall loudness of snoring with score of 0 meaning no snoring and 10 meaning extreme snoring

SECONDARY OUTCOMES:
Change in Epworth Sleepiness Scale | At 2 weeks, at 6 weeks and at 6 months
  Seld-reported subjective score that evaluates the presence of hypersomnolence. Score out of 24 with 0 meaning no hypersomnolence and 24 extreme hypersomnolence

CONTACTS AND LOCATIONS:
Locations (1):
- Neus-, keel- en oorziekten, gelaats- en halschirurgie AZ Delta, Roeselare, Belgium

IPD SHARING:
Plan to Share IPD: No